CLINICAL TRIAL: NCT03553485
Title: Effects of Transcutaneous Auricular Vagal Nerve Stimulation on Radiotherapy-induced Inflammation and Prognosis of Patients With Lung Cancer
Brief Title: Effects of VNS on RT-induced Inflammation and Prognosis of Patients With NSCLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Kom Op Tegen Kanker (Other)
Responsible Party: Principal Investigator, Reijmen Eva, Principal Investigator, Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1.0_09/01/2018
Record Dates: First submitted 2018-05-11; First posted 2018-06-12 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Lung Cancer, Non-small Cell
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- taVNS (Experimental): Treatment will be carried out twice a day (once before the RT session and 8h later) during 7 weeks. Each treatment takes 30 minutes.
  Interventions: Device: Transcutaneous vagus nerve stimulation; Radiation: Radiotherapy
- Control (Sham Comparator): Treatment will be carried out twice a day (once before the RT session and 8h later) during 7 weeks. Each treatment takes 30 minutes.
  Interventions: Device: Sham; Radiation: Radiotherapy

INTERVENTIONS:
Device: Transcutaneous vagus nerve stimulation — The transcutaneous auricular vagus nerve stimulator Parasym consists of a stimulation unit and a dedicated ear electrode. The stimulation unit, having approximately the size of a common mobile phone, sends out the electrical impulses. It is connected with the ear electrode, which patients wear like an earphone. The patient can regulate and adapt the intensity of the stimulation (current intensity) according to his/her individual sensitivity, which can vary from day to day or even over the period of the therapy.
  Arms: taVNS
Device: Sham — Sham Earclip electrodes are electrodes that appear identical to functioning electrodes, however do not deliver any stimulation due to removed wiring.
  Arms: Control
Radiation: Radiotherapy — Standard treatment for included patients

SUMMARY:
Lung cancer (LC) remains a leading cause of death among cancers worldwide. Though radiotherapy is one of the most frequently used treatments, it increases side-effects (pain, fatigue) and inflammation, possibly leading to further tumorigenesis of surviving cancer cells. The purpose of this study is to test the effects of transcutaneous auricular VNS vagal nerve stimulation (taVNS), known to reduce inflammation, on radiotherapy-induced inflammation and other side-effects in LC patients undergoing radiotherapy.

In this feasibility study 12 patients with NSCLC stage III (A/B) receiving radiotherapy will be enrolled. Our primary endpoint is the effect of vagus nerve stimulation (VNS) on inflammatory levels (such as CRP and cytokines), immunological factors (neutrophils, monocytes, lymphocytes) and the tumor marker CEA. Our secondary endpoint is the psychological well-being and quality of life of the patients during their radiotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old
* Patients with non-small cell lung cancer stage III (A or B)
* Patients receiving radiotherapy or chemoradiotherapy
* Patients with an HRV < 70 msec

Exclusion Criteria:

* Patients with an active implantable medical device, such as a pacemaker, hearing aid implant or any other implanted electronic device
* Patients with an implanted or wearable defibrillator.
* Patients with myocardial disease
* Patients with arrhythmias
* Patients with an implanted metallic or electronic device in their head.
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-08-08 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Cancer prognosis: tumor marker | 7 weeks
  CEA (µg/mL)
Cancer prognosis: inflammatory level | 7 weeks
  CRP (mg/mL)
Cancer prognosis: inflammatory level | 7 weeks
  cytokines: IL1, IL2, IL6 and IL8 (pg/mL)
Cancer prognosis: immunological factors | 7 weeks
  neutrophil count (x10³/mm³)

SECONDARY OUTCOMES:
Health related Quality of Life | 7 weeks
  To assess the psychological well-being and quality of life of the patients during their radiotherapy treatment the EORTC QLQ-C30 questionnaire will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Reijmen, Dra, Principal Investigator — VUB
Locations (1):
- UZ Brussels, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No